CLINICAL TRIAL: NCT03879330
Title: NIRS Directed Optimal Cerebral Perfusion Pressure in Aneurysmal Subarachnoid Hemorrhage Patients: A Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018101083
Record Dates: First submitted 2019-03-06; First posted 2019-03-18 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2018-10

CONDITIONS: The Time for Determine CPPopt

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NIRS monitoring — aSAH patients will be given continuous NIRS and blood pressure monitoring at same time. The correlation curve between the brain oxygenation index or the brain hemoglobin index (ORI/THx) and the blood pressure will be obtained through continuous monitoring of 4 hours. According to the correlation curve, the optimal blood pressure will be determined which provides the optimal CPP.

SUMMARY:
Neurologic dysfunction is common in aneurysmal subarachnoid hemorrhage (aSAH) patients. As we know, after the initial injury, secondary insults including poor cerebral perfusion are main contributors to poor outcome and their early detection and amelioration are keystone to neurocritical care. Nonetheless, the guidelines for blood pressure management still recommend a single target blood pressure for critically ill patients: the Brain Trauma Foundation (BTF) guidelines recommend maintaining CPP between 60 and 70 mmHg; Some guidelines recognize that patients with a history of hypertension may require a higher MAP. However, these guidelines do not currently recommend cerebral autoregulation-guided therapy and leave many unanswered questions. Cerebral autoregulation is the mechanism that maintains cerebral blood supply, hence CBF approximately constant despite changes in MAP or, more precisely, despite changes in CPP. Maintaining blood pressure within the cerebral blood flow (CBF) autoregulation range (termed "optimal MAP") is associated with improved outcomes for patients. The observational data suggests that management of patients above or below CPPopt 5mmHg is associated with better outcomes and mortality than the other greater variation range. The most commonly used method for monitoring dynamic cerebrovascular reactivity is the pressure reactivity index (PRx) that uses ICP as a surrogate for CBV. However, assessing the PRx requires invasive ICP monitoring which limits its application in many clinical areas. Alternatively, in the absence of invasive intracranial pressure monitoring to determine CPP, a continuous autoregulation monitoring can be accomplished by the continuous correlation between transcranial Doppler (TCD)-measured CBF velocity of the middle cerebral artery and the mean arterial blood pressure (termed mean velocity index or Mx). Mx is a validated index of cerebral autoregulation based on measures of cerebral perfusion pressure and mean flow velocity on transcranial doppler but is impractical for longer-term monitoring and requires system training, the results are operator-dependent. Near-infrared spectroscopy (NIRS) measurements is another alternative for real-time autoregulation monitoring in the form of a Tissue Oxygenation Index. In contrast to TCD, the NIRS sensors are very easy to apply (the probes attach to the forehead with self-adhesive pads) and do not require frequent calibration making them more suitable for long-term monitoring. Therefore, in this study, Patients in the intervention group will be monitored by continuous NIRS and invasive blood pressure monitoring. The correlation curve between ORI/THx and blood pressure will be obtained through continuous monitoring of 2 hours. According to the correlation curve, the optimal blood pressure which provides the optimal CPP will be determined. Then the optimal blood pressure which CPP is within 5 mmHg of CPPopt will be maintained as the target of blood pressure management for the intervention group during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Admitted to ICU because of aSAH (Hunt & Hess classification≥ 3).
3. Predicted to stay in ICU ≥ 24 hours

Exclusion Criteria:

1. Unable to perform NIRS monitoring because of anatomic factors: such as forehead skin damage, intracranial gas accumulation, severe edema of monitoring sites;
2. Patients with severe organ failure: such as poorly controlled chronic hypertension, chronic renal failure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (Age ≥ 18 years) aneurysmal subarachnoid hemorrhage patients (Hunt & Hess classification≥ 3) who admitted to ICU and predicted to stay in ICU ≥ 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimal CPP | 16 hours
  the minimal time that CPPopt can be determined by the correlation curve between the brain oxygenation index or the brain hemoglobin index (ORI/THx) and the blood pressure.

IPD SHARING:
Plan to Share IPD: Undecided